CLINICAL TRIAL: NCT01124123
Title: Study to Assess Oral Bioavailability of Bilastine (Estudio de Biodisponibilidad Oral de Bilastina)
Brief Title: Oral Bioavailability of Bilastine
Acronym: BIOBI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Faes Farma, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: BILA 2909/BA; 2010-019049-25 (EudraCT Number)
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Oral bioavailability; absorption; AUC; Bioequivalence; Bioavailability study
MeSH Terms: interventions — bilastine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bilastine 20 mg (Experimental): Single dose 20 mg bilastine oral tablet. Test drug
  Interventions: Drug: Bilastine
- Bilastine 10 mg (Active Comparator): Single dose 10 mg Bilastine endovenous. Control drug
  Interventions: Drug: Bilastine

INTERVENTIONS:
Drug: Bilastine — 20 mg oral tablet
  Arms: Bilastine 20 mg
Drug: Bilastine — 10 mg endovenous bilastine
  Arms: Bilastine 10 mg

SUMMARY:
The purpose of this study is to assess the absolute bioavailability of an oral bilastine formulation (test drug) compared to the endovenous administration of an IV bilastine formulation (control drug) in healthy volunteers.

DETAILED DESCRIPTION:
Single centre, open label, cross-over, randomised, controlled, single dose study. The primary endpoint is the determination of plasma concentrations versus time (17 samples per subject at various time intervals after dosing) in order to assess the oral bioavailability of bilastine in healthy volunteers. Therefore the primary pharmacokinetic variable will be the area under the plasma concentration versus time curve from time zero to infinity (AUC 0-∞). Additionally the following pharmacokinetic variables will also be assessed: Cmax, AUC 0-t, tmax, Ae, Clr, t1/2. Additional objectives are to describe the safety and tolerability of a single administration of oral and endovenous bilastine in healthy volunteers.

Twelve healthy volunteers will be included. Each volunteer will take in random order one single dose of 20 mg oral bilastine and 10 mg IV bilastine with a minimum washout period of 14 days between them.

Bilastine plasma concentrations will be measured using a liquid chromatography/mass mass spectrometry (LC/MS/MS) micro method

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers of either sex aged from ≥ 18 to ≤ 35 years of age.
* Body mass index between 19 and 29 Kg/m2.
* Non smokers.
* Judged to be in general good health based on medical history, physical examination and clinical laboratory tests.
* Able to communicate well with the investigator and to comply with the requirements of the entire study.
* Provision of written informed consent to participate.

Exclusion Criteria:

* Pregnant or breast-feeding women or with a positive pregnancy test. Subjects who do not agree to use an adequate method of contraception during the study.
* Intake of another investigational medication in another clinical study within 4 months prior to the first study drug intake.
* Regular use of any prescribed medication including medicinal herbs or OTC medication within 4 weeks of dosing.
* A QTc> 430 ms in males and a QTc> 450 ms in females. A HR <55 bpm.
* Existence of any surgical or medical condition which, in the judgement of the investigator, might interfere with the absorption, distribution, metabolism or excretion of the IMP.
* Known allergy/hypersensitivity to the study drug or its inactive ingredients.
* Any clinical conditions or circumstances that in the opinion of the investigator would make the subject unsuitable for the study (e.g., hepatic impairment, renal impairment, mental impairment, cardiac disease).
* Presence of hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab) or HIV 1 or HIV 2 antibodies at screening.
* Subjects who have taken metabolic or transporter inducers/inhibitors during the 3 months prior to inclusion in the study.
* Donation or loss of greater than 200 mL of blood within 12 weeks before entry to the study.
* Blood transfusion within the prior 6 months to inclusion.
* Ingestion of citrus fruits and cranberries or any fruit juice within 7 days prior to first dose of study medication.
* Known current alcohol or drug abuse.
* Excessive consumption of xanthine containing foods or drinks.
* Mentally disabled subjects or subjects who by official order have been institutionalised must be excluded from participation.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
The area under the plasma concentration versus time curve from time zero to infinity (AUC 0-∞ ). | 17 blood draws performed at: 0,25 - 0,5- 0,75 - 1 - 1,25 - 1,5 - 1,75 - 2 - 2,5 - 3 - 4 - 5 - 7 - 12 - 24 - 48 and 72 hours post administration.
  Bilastine bioavailability will be obtained from the oral AUC 0-∞ / endovenous AUC 0-∞ quotient.

SECONDARY OUTCOMES:
Additional pharmacokinetic variables: Cmax, AUC 0-t, tmax, Ae, CLr and t ½ | 17 blood draws and urine collection during 72 hours post administration
  * Cmax: Maximum plasma concentration; the highest concentration observed during a dosage interval
  * tmax: The time that Cmax was observed
  * AUC 0-t: The area under the plasma concentration versus time curve from time zero to the last time point
  * Ae: amount of accumulated unaltered drug in urine till the last time point
  * Clr: Renal clearance
  * t ½: Elimination halflife
Safety and tolerability of a single dose administration of oral and endovenous bilastine | A last Follow up visit will be performed 7 days after last drug intake
  Safety will be assessed during the study by monitoring adverse events (AEs), clinical laboratory test results (urinalysis, blood chemistry, and haematology), vital signs (including blood pressure, respiration, temperature, and heart rate, supine and standing), electrocardiogram (ECG) results, and abnormal findings upon physical examination.

CONTACTS AND LOCATIONS:
Overall Officials: Belen Sadaba, MD, Principal Investigator — Unidad de Investigacion Clinica. Clinica Universidad Navarra (CUN)
Locations (1):
- Unidad de Investigacion Clinica. Clinica Universidad de Navarra, Pamplona, Navarre, Spain

REFERENCES:
- [Background] Jauregizar N, de la Fuente L, Lucero ML, Sologuren A, Leal N, Rodriguez M. Pharmacokinetic-pharmacodynamic modelling of the antihistaminic (H1) effect of bilastine. Clin Pharmacokinet. 2009;48(8):543-54. doi: 10.2165/11317180-000000000-00000. PMID 19705924
- [Background] Lucero ML, Gonzalo A, Ganza A, Leal N, Soengas I, Ioja E, Gedey S, Jahic M, Bednarczyk D. Interactions of bilastine, a new oral H(1) antihistamine, with human transporter systems. Drug Chem Toxicol. 2012 Jun;35 Suppl 1:8-17. doi: 10.3109/01480545.2012.682653. PMID 22616811
- [Derived] Sadaba B, Gomez-Guiu A, Azanza JR, Ortega I, Valiente R. Oral availability of bilastine. Clin Drug Investig. 2013 May;33(5):375-81. doi: 10.1007/s40261-013-0076-y. PMID 23529786
- See also: Clinical Trials and Medical Research page. Clinica Universidad Navarra (CUN) — http://www.cun.es/nc/la-clinica/investigacion/ensayos-clinicos/
- See also: Clinical Pharmacology Department. Clinica Universidad Navarra (CUN) — http://www.cun.es/la-clinica/servicios-medicos/farmacologia/